CLINICAL TRIAL: NCT03553901
Title: The Effect of Acupressure (GB30) on Ventrogluteal Intramuscular Injection Pain - A Crossover Randomized Single-blind Study
Brief Title: The Effect of Acupressure (GB30) on Ventrogluteal Intramuscular Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sultan Abdulhamid
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Acute Pain; Injection; Needle Phobia
MeSH Terms: conditions — Acute Pain | interventions — Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure (Experimental): Acupressure is applied before injection
  Interventions: Procedure: Acupressure
- Control group (No Intervention): acupressure is not applied before injection

INTERVENTIONS:
Procedure: Acupressure — Acupressure was performed before the injection onto GB30 point
  Arms: Acupressure

SUMMARY:
Acupressure is an ancient manual therapy which fingers are used to press key points on the body. These points are the same with acupuncture points but in contrast to acupuncture, acupressure uses gentle but firm pressure with fingers and hands. The purpose of this study is to investigate effect of acupressure onto GB30 poin for ventrogluteal intramuscular injection pain.The study was designed as a prospective, single-blind, crossover study. The study included 72 volunteer students attending Faculty of Health Sciences, Nursing Department.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18.5 to 29.9kg/m2
* Voluntariness

Exclusion Criteria:

* history of IM injection within 2 weeks

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Assessment of pain during intramuscular injection with 10 cm VAS (Visual Analog Scale) | 2 minutes
  Assessment of pain during intramuscular injection will be marked on 10 cm VAS scale 0-10 ( 0:no pain 10:Worst possible pain ) by the patient and will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan inangil, Study Director — Sultan Abdulhamid Han

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Suhrabi Z, Taghinejad H. Effect of acupressure (UB32) on pain intensity in intramuscular injections. Iran J Nurs Midwifery Res. 2014 Jan;19(1):24-7. PMID 24554956
- [Background] Hosseinabadi R, Biranvand S, Pournia Y, Anbari K. The Effect of Acupressure on Pain and Anxiety Caused by Venipuncture. J Infus Nurs. 2015 Nov-Dec;38(6):397-405. doi: 10.1097/NAN.0000000000000065. PMID 26536327
- [Background] Chung JW, Ng WM, Wong TK. An experimental study on the use of manual pressure to reduce pain in intramuscular injections. J Clin Nurs. 2002 Jul;11(4):457-61. doi: 10.1046/j.1365-2702.2002.00645.x. PMID 12100641